CLINICAL TRIAL: NCT01972594
Title: A 12 Week Pedometer Based Walking Intervention to Enhance Physical Activity Performance Following Total Hip Replacement-A Pilot Study
Brief Title: Pedometer Based Intervention After Total Hip Replacement-A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ben Stansfield (Other)
Collaborators: Golden Jubilee National Hospital (Other Government)
Responsible Party: Sponsor-Investigator, Ben Stansfield, Academic Supervisor to the Chief Investigator of the Study, Glasgow Caledonian University
Organization: Glasgow Caledonian University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: GCU_ALARG_AJ_002
Record Dates: First submitted 2013-10-16; First posted 2013-10-30 (Estimated); Last update posted 2015-03-13 (Estimated); Status verified 2015-03

CONDITIONS: Osteoarthritis of Hip
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group. (No Intervention): Natural progession based on Step count is recorded with a pedometer for 12 weeks.
- Targeted protocol with Pedometer (Experimental): A step based targeted protocol is given along with a pedometer for 12 weeks post surgery.
  Interventions: Procedure: Targetted protocol with pedometer; Device: Accelerometer(ActivPAL)

INTERVENTIONS:
Procedure: Targetted protocol with pedometer — 12 week protocol based on targetted steps are given to the patient along with a pedometer.
  Arms: Targeted protocol with Pedometer
Device: Accelerometer(ActivPAL)
  Arms: Targeted protocol with Pedometer

SUMMARY:
Total hip replacement is designed to alleviate pain, reduce disability and improve function and physical activity levels. Whilst pain, disability and function are often measured following surgery, actual physical activity is not. The aim of rehabilitation after total hip replacement would be to obtain optimal strength and range of movement at the hip along with cumulative endurance and balance. It is taken for granted that, once function is restored, the patient returns to physical activity levels associated with good health. In a previous study conducted by the same team it was observed that patients, at the end of 3 months after hip surgery, do not reach the levels of physical activity which are proven to be beneficial for health. Physiotherapy plays an important role in improving function and increasing levels of Physical activity in total hip replacement patients, but there is limited literature to substantiate this claim. There is a need to enhance levels of physical activity in patient after total hip replacement towards levels that are associated with good health. This study aims to demonstrate a method of enhancing physical activity levels after total hip replacement using a pedometer based intervention over a period of 3 months. Patients will follow a customized progressive stepping activity schedule aimed at establishing levels of physical activity that are associated with good health. To fully understand recovery patterns subjective and objective measures of strength of the hip muscles, range of motion at the hip, overall endurance, balance and speed of walking of the patient will be assessed. Questionnaires will be utilized to assess quality of life both before and after total hip surgery. The physical activity levels of the patient will be measured with a physical activity monitor. This study will be completed at the Golden Jubilee National Hospital at Glasgow.

DETAILED DESCRIPTION:
Physical activity can be defined as the time spent engaging in non-sedentary behaviour. This would include sit to stand episodes, periods spent upright and periods spent stepping. Physical activity can be considered as purposeful free living activity with major health benefits. According to the World health organisation, Physical activity is defined as any bodily movement produced by skeletal muscles that requires energy expenditure. Physical inactivity has been identified as the fourth leading risk factor for global mortality causing an estimated 3.2 million deaths globally. Improvement in Physical activity levels has a direct and indirect add-on effect in reducing various comorbidities which may or may not exist in a patient including cardiac diseases, stroke, diabetes and osteoporosis. These facts can also be applied to orthopedically challenged individuals undergoing total hip replacement or recovering from it.

Total hip replacement (THR) or total hip arthroplasty (THA) is one of the most common orthopaedic surgeries performed and has been termed as the "operation of the century". It has been suggested that impairment and physical limitations persisted in the long-term following a THR, even in the absence of pain, with reduced muscle strength, postural stability and flexibility. These factors would indirectly affect the physical activity levels of a patient which neutralizes one of the purposes of the total hip replacement. Reduction in the ability to be physically active is one of the reasons a patient undergoes a total hip replacement, others being pain and disability. One of the goals of the orthopaedic surgeon is to bring a patient back to an acceptable level of physical function and activity, post-surgery. This depends on both compliance with rehabilitation programmes and ability of the patient. Previously is has been found that there is only a small increase in patients' actual physical activity at post THR surgery, possibly due to the lifestyle changes adopted by the patients to manage their condition prior to undergoing surgical intervention.

Physiotherapy is the mainstay of treatment for post-operative total hip replacements as it attempts to address the issues of impairment, disability and function. The use of physiotherapy as an intervention either before or after surgery has been investigated, with evidence to suggest that there are benefits to outcome. Post-operative physical training which includes physiotherapy is beneficial to patients with a THR, even if they have co-morbidities. It has been proposed that early and late post-operative protocols should include treadmill training, resistance training for the quadriceps muscles, arm interval exercise training with weight bearing exercises and eccentric training of the hip abductors. These protocols appeared to provide benefits for the participants, increasing strength, endurance and balance. However, they may not be applicable clinically in the current socio economic scenario. There is a need for effective and simple protocols which can be implemented across a range of patient groups in a cost effective manner.

After undergoing the required rehabilitation programs post major surgery there appears to be a gap in the literature available as to the improvement and sustenance of physical activity levels. If physical activity is a key component of a healthy life style then its promotion and monitoring would enhance and inform the rehabilitation process. The promotion of physical activity has been successful in populations using pedometers as motivational tools. Whilst, these interventions have been implemented widely there is limited evidence specifically in populations following orthopaedic surgery. Perhaps this is because recovery to 'healthy' levels of activity has not been seen as an important objective of the rehabilitation process and simple functional recovery is all that has been targeted.

'Participation' as defined within the World Health Organisation's International Classification of Functioning, Disability and Health classification tree is concerned with the free-living activity of individuals. The measurement of participation is difficult, except through a questionnaire based approach. To overcome the subjective nature of questionnaires, body worn monitors have been developed that allow the quantification of aspects of posture and stepping activity. Whilst the measurement of ability goes some way towards understanding the positive benefits of hip replacement as an intervention, knowledge of free-living activity would considerably extend the clinician/health professional understanding of the patient's recovery following the operation. Conventional tools for assessing participation include questionnaires such as the SF36, WOMAC, UCLA, Hip dysfunction and Osteoarthritis Outcome Score, Harris Hip Score and the Oxford Hip Score. Objective measurement of physical activity (e.g. using body worn monitors) removes the subjectivity of questionnaires. There is clearly a cost and time implication for the use of monitoring devices, so it is important that they provide additional, valuable information on free-living physical activity in comparison to quick to implement and readily accessible questionnaires.

Modern pedometers are small, user friendly and relatively inexpensive (approximately £20), providing a suitable tool for wide spread use. Pedometers can be used both as a means of providing motivation for enhanced physical activity and as a monitoring device to quantify this activity. The use of such devices within interventions to enhance physical activity must be based on evidence of effectiveness. It has been established that the number of steps achieved in a day can be used to categorise physical activity levels. The 'step defined lifestyle index' categorises individuals taking less than 5000 steps/day as sedentary, 5000-7499 steps/ day as low active lifestyle and more than 7500 steps/day as physically active. Those individuals meeting the 7500+ threshold appear to meet the moderate to vigorous physical activity recommendations for health. It is also suggested that achieving 7000- 8000 steps per day Is associated with achieving 30 minutes per day of moderate to vigorous physical activity. To gain an understanding of the significance of the stepping guidelines, it has been established that 3000 accumulated purposeful steps per day equate to 30 minutes of moderate physical activity, which is the recommended daily physical activity quotient for good health. These recommendations can be used as targets, not only for healthy individuals but also for others including orthopedically challenged patients recovering from surgery.

In a previous, observational study ( the research team have followed total hip replacement patients from before surgery to 3 months after surgery. Over this period the relationship between physical activity performance and aspects of ability and activity limitation was measured under laboratory/clinical conditions and free-living activity was recorded using a body worn activity monitor. This observational study revealed a number of facts about the recovery process post-surgery:

1. At 3 month post-surgery, pain was generally absent and there was an improvement in hip strength and aerobic endurance. However, patients' hip strength and aerobic endurance, at 3 months after surgery, were observed to be far below the reference values of age and sex matched healthy individuals.
2. Patients who were relatively active before undergoing total hip replacement, remained relatively active at the 3 month follow-up.
3. The average number of steps taken by the patients before surgery was around 5200 steps per day and after surgery at the 3 month follow-up was approximately 5800 steps per day.
4. However, 46 % of patients achieving less than 5000 steps per day at 3 months post-surgery.
5. There was a direct relationship between the endurance of a patient and the physical activity levels achieved by the patient at 3 month follow up.
6. It was also noted that the average time spent by the subjects in a sedentary position, i.e. sitting or lying, had minimally reduced per day from pre-surgery to the 3 month follow-up.

Whilst some of the patients recovered to physical activity levels that are associated with good health, a large proportion did not. The need for a strategy to increase physical activity within this patient group is clear. Previous examples of successful pedometer based interventions motivate the current study which will aim to improve physical activity performance towards levels that are recognised to be health sustaining. The outcome measures used within the observational study will be repeated to allow direct comparison between study groups.

The purpose of the proposed study is to investigate outcomes of a pedometer based intervention to improve physical activity levels and to examine if there could be a crossover effect of changes in stepping activity to hip strength and endurance following hip replacement surgery.

The Chief investigator has undergone training in Good clinical practice and governance and has the experience of doing hospital based research.

ELIGIBILITY:
Inclusion Criteria:

* Primary total hip replacement
* Age group between 60-80 years old.
* Able to give informed consent
* Able to return for follow-up
* Able to read and understand English and follow verbal and visual instructions

Exclusion Criteria:

Bilateral total hip replacements

* Either hip or knee replacement in the last 12 months
* Severe locomotor limitation due to cardio-respiratory dysfunction
* Severe locomotor disorder due to central or peripheral nervous system deficits
* Severe locomotor limitation due to spinal condition
* Severe locomotor limitation due to musculoskeletal disabilities
* Diagnosed terminal

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-01; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Change in Physical Activity following Hip Replacement. | pre-operative,Immediate post -operative,1st week post operative and 3 months post operative.
  Free-living physical activity performance will be recorded using an Accelerometer(ActivPAL).A small CE marked physical activity monitor, ActivPAL (PAL Technologies Ltd. Glasgow, UK) will be attached to the anterior thigh (of the non-operated leg) using a water proof surgical dressing material. This monitor, with proven validity is 50mm x 35mm x 7mm and weighs 30g. The fixing with the dressing allows it to be worn continually without affecting any patient activity such as washing / showering etc. This remains in place for the duration of the recording. It can record date for up to 7 days. The time spent upright, time spent stepping and the numbers of steps taken are recorded continuously over multiday periods. The intervention group will be encouraged to increase their physical activity levels. This will be based on a measure of stepping activity and a pedometer will act as a guideline for how many steps are required per day.

CONTACTS AND LOCATIONS:
Locations (1):
- Golden Jubilee National Hospital, Glasgow,Scotland, United Kingdom

REFERENCES:
- See also: Golden Jubilee national Hospital Website. — http://www.nhsgoldenjubilee.co.uk/